CLINICAL TRIAL: NCT04483427
Title: Multimodal Postoperative Analgesia Using Accufuser for Multilevel Surgery for Obstructive Sleep Apnea (OSA)
Brief Title: Multimodal Postoperative Analgesia Following OSA Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bahaa Mohammed Refaie (Other)
Responsible Party: Sponsor-Investigator, Bahaa Mohammed Refaie, Lecturer of anesthesia and ICU, Sohag University
Organization: Sohag University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1984
Record Dates: First submitted 2020-07-16; First posted 2020-07-23 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Nalbuphine; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OSA patients after multilevel surgery (Experimental)
  Interventions: Combination Product: Nalbuphine, ketorolac, accufuser

INTERVENTIONS:
Combination Product: Nalbuphine, ketorolac, accufuser — multimodal analgesic regimen consisting of nalbuphine combined with ketorolac using IV continuous infusion silicon device (Accufuser)

SUMMARY:
Assessment of the clinical efficacy and adverse effects of multimodal analgesic regimen consisting of nalbuphine combined with ketorolac using IV continuous infusion silicon device (Accufuser) for postoperative analgesia following multilevel OSA surgeries

ELIGIBILITY:
Inclusion Criteria:

* physical status of American Society of Anesthesiologists (ASA) II
* age between 30 - 50 years
* OSA patients diagnosed by polysomnography and stop-bang questionnaire
* enrolled for multilevel OSA surgery

Exclusion Criteria:

* history of allergy to the study drugs
* history of hepatic, cardiopulmonary or renal disease
* history of any chronic pain on medication
* history of substance abuse
* psychiatric disorder
* lack of patient cooperation.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Assessment will be carried out at zero time (time to shift to PACU) .
  visual analog pain score
Postoperative pain | Assessment will be carried out 6 hours postoperatively
  Visual analog pain score
Postoperative pain | Assessment will be carried out 12 hours postoperatively
  Visual analog pain score
Postoperative pain | Assessment will be carried out 18 hours postoperatively
  Visual analog pain score
Postoperative pain | Assessment will be carried out 24 hours postoperatively
  Visual analog pain score
Postoperative pain | Assessment will be carried out 30 hours postoperatively
  Visual analog pain score
Postoperative pain | Assessment will be carried out 36 hours postoperatively
  Visual analog pain score
Postoperative pain | Assessment will be carried out 42 hours postoperatively
  Visual analog pain score
Postoperative pain | Assessment will be carried out 48 hours postoperatively
  Visual analog pain score

SECONDARY OUTCOMES:
Sedation level | Zero time ( time to shift to PACU)
  Ramsey sedation scale
Sedation level | 6 hours postoperatively
  Ramsey sedation scale
Sedation level | 12 hours postoperatively
  Ramsey Sedation Scale
Sedation level | 18 hours postoperatively
  Ramsey Sedation Scale
Sedation level | 24 hours postoperatively
  Ramsey Sedation Scale
Sedation level | 30 hours postoperatively
  Ramsey Sedation scale
Sedation level | 36 hours postoperatively
  Ramsey Sedation Scale
Sedation level | 42 hours postoperatively
  Ramsey Sedation Scale
Sedation level | 48 hours postoperatively
  Ramsey Sedation Ramsey Sedation Scale
incidence of adverse effects | Zero time ( time to shift to PACU)
  hypoxia, nausea, vomiting, itching
incidence of adverse effects | 6 hours postoperatively
  hypoxia, nausea, vomiting, itching
incidence of adverse effects | 12 hours postoperatively
  hypoxia, nausea, vomiting, itching
incidence of adverse effects | 18 hours postoperatively
  hypoxia, nausea, vomiting, itching
incidence of adverse effects | 24 hours postoperatively
  hypoxia, nausea, vomiting, itching
incidence of adverse effects | 30 hours postoperatively
  hypoxia, nausea, vomiting, itching
incidence of adverse effects | 36 hours postoperatively
  hypoxia, nausea, vomiting, itching
incidence of adverse effects | 42 hours postoperatively
  hypoxia, nausea, vomiting, itching
incidence of adverse effects | 48 hours postoperatively
  hypoxia, nausea, vomiting, itching

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa M Refaie, MD, Principal Investigator — Lecturer of anesthesia and ICU sohag university; Mohammed E Ahmed, MD, Study Director — Lecturer of ENT sohag university; A M Elhalwagy, MD, Study Chair — Consultant of pain medicine
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided